CLINICAL TRIAL: NCT01672762
Title: Phase III Study of ASP1941 -A Phase III, Open-Label, Uncontrolled, Monotherapy Study to Assess the Long-term Safety, Tolerability and Efficacy of ASP1941 in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate Long-term Safety and Efficacy of ASP1941 in Diabetes Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1941-CL-0122
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: glucose excretion; ipragliflozin; hypoglycemic agents; serum Insulin; diabetes mellitus; blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ipragliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP1941 group (Experimental): oral
  Interventions: Drug: ipragliflozin

INTERVENTIONS:
Drug: ipragliflozin — oral
  Other Names: ASP1941

SUMMARY:
This study is to evaluate safety and efficacy of ASP1941 after 24 week administration to diabetic patients.

DETAILED DESCRIPTION:
Subjects will undergo the 6-week screening period before entering the 24-week treatment period and will receive ASP1941 before breakfast during the treatment period. All subjects will be followed for 4 weeks after study treatment is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patients
* Subject is only on a diet and exercise program or has received a single antihyperglycemic agent or two antihyperglycemic agents (excluding insulin) with low dose (≤50% of the maximum dose of each recommended dosage)
* Subject has a HbA1c value (JDS value) between 6.5% and 9.5% and the difference of HbA1c values (JDS value) within ± 1.0%
* BMI 20.0 - 45.0 kg/m2

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* Subject has received insulin within 12 weeks (84 days) before the study
* Subject has proliferative diabetic retinopathy
* Subject has a history of clinically significant renal disease such as renovascular occlusive disease, nephrectomy and/or renal transplant
* Subject with obvious dysuria caused by a neurogenic bladder or a benign prostatic hypertrophy
* Subject has a history of cerebral vascular attack, unstable angina, myocardial infarction, vascular intervention, and heart disease (NYHA Class III-IV) within 12 weeks (84 days). Subject has heart disease, cerebral vascular disease which, in the opinion of the principal investigator or the sub-investigator, may interfere with treatment or evaluation of safety of this study.
* Female subject who is currently pregnant or lactating, or who is possibly pregnant
* Male and pre-menopausal Female subject who cannot use an appropriate contraception during the study
* Subject has a history of treatment with ASP1941
* Subject has participated in another clinical study, post marketing study, or medical equipment study within 12 weeks (84 days) before providing written informed consent, or who is currently participating in any of those studies
* Subject has a serum creatinine value higher than upper limit of normal range
* Subject has a urinary microalbumin/ urinary creatinine ratio > 300 mg/g in urinalysis
* Subject has uncontrolled severe hypertension (subject whose systolic blood pressure is > 170 mmHg or diastolic blood pressure of > 95 mmHg measured in a sitting position after 5 minutes of rest
* Subject who is judged inappropriate for enrollment into the study by the principal investigator or the sub-investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2012-05-25 (Actual); Primary Completion 2013-04-13 (Actual); Study Completion 2013-04-13 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Before and at 4-, 8-, 12-, 16-, 20- and 24-week

SECONDARY OUTCOMES:
Change in fasting plasma glucose | Before and at 4-, 8-, 12-, 16-, 20- and 24-week
Change in fasting serum insulin | Before and at 4-, 8-, 12-, 16-, 20- and 24-week
Change in waist circumference | Before and at 4-, 8-, 12-, 16-, 20- and 24-week
Change in body weight | Before and at 4-, 8-, 12-, 16-, 20- and 24-week
Change in urine glucose | Before and at 4-, 8-, 12-, 16-, 20- and 24-week
Safety assessed by the incidence of adverse events, vital signs, lab-tests and 12-lead ECGs | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=107